CLINICAL TRIAL: NCT00681681
Title: Sex Differences in Vascular Markers of Stroke Risk
Acronym: SAVVY
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: K02NS058760 (NIH); IRB00004014 (Other: Wake Forest University Health Sciences); K02NS058760-01A1 (NIH)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2014-12

CONDITIONS: Stroke
Keywords: stroke; vascular marker; stroke risk; risk factors; sex differences
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA and DNA samples collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Men and women with 1 or more cardiovascular risk factors

SUMMARY:
The purposes of this study are to quantify and compare vascular function in men and women, and to determine the effect of age, race-ethnicity, cardiovascular risk factors, biological markers and hormonal markers on vascular measures to establish gender-specific models.

DETAILED DESCRIPTION:
Men and women with stroke have different risk factor profiles. Women tend to develop stroke risk factors, subclinical disease, and have vascular events following menopause, presumably related to the depletion of estrogen. Men, however, tend to develop vascular disease at a younger age. Sex differences in subclinical disease are poorly understood. Identification of subclinical disease could lead to more aggressive interventions to prevent stroke and other vascular events.

The objectives of this study are to quantify and compare vascular function in men and women by measuring carotid atherosclerosis, endothelial dysfunction, and ankle-brachial index and then to determine the effect of age, race-ethnicity, cardiovascular risk factors, biological markers and hormonal markers on these vascular measures to determine gender-specific models. The aims of this project are to determine if middle-aged men and women at risk for stroke have differences in functional and structural vascular assessments, and to develop comprehensive vascular health profiles in men and women.

In this trial, researchers will use a cross-sectional design to study gender differences in vascular functions and other vascular risk factors in 150 women and 100 men with 1 or more cardiovascular risk factors but without evidence of stroke, heart disease, or peripheral vascular disease. Participants will be divided in two age groups: 45 to 54 and 55 to 64 and will be followed for two years for vascular outcomes, such as stroke, transient ischemic attack or TIA, or acute coronary syndromes.

Information from this study will help develop a comprehensive gender-specific model of subclinical disease, discover novel biological and vascular markers for stroke, and provide critical data to be used in future studies aimed at slowing progression of vascular dysfunction and preventing stroke.

ELIGIBILITY:
Inclusion Criteria:

One or more cardiovascular risk factors

* non-insulin dependent diabetes
* hypertension
* hyperlipidemia
* metabolic syndrome, (NCEP ATPIII criteria)
* tobacco smoking

Exclusion Criteria:

* history of prior stroke (ischemic or hemorrhagic)
* TIA
* known carotid stenosis
* peripheral vascular disease
* coronary heart disease
* venous thromboembolism
* polycystic ovarian syndrome,
* morbid obesity (BMI > 45 kg/m2)
* women using hormone therapy (hormone replacement, contraceptive pills or patches)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from primary care clinics, which may include internal medicine, family practice, and obstetrics/gynecology within the Wake Forest University health system.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2008-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Carotid intimal medial thickness (IMT) and 10-year cardiovascular risk assessment. The primary analysis will focus on gender differences. | 3 years

SECONDARY OUTCOMES:
Brachial artery flow mediated dilation (BAFMD) and ankle-brachial index (ABI) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Bushnell, MD, Principal Investigator — Associate Professor, Department of Neurology, Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States